CLINICAL TRIAL: NCT06263751
Title: NutriConnect: Enhancing Health and Food Security Through Sustainable Solutions and Partnerships
Brief Title: Comparing the Effectiveness of Two Produce Prescription Approaches On Fruit and Vegetable Intake and Food Security, While Exploring Implementation Outcomes Such as Reach, Implementation, Sustainability, and Cost
Acronym: NutriConnect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Schnuck Markets, Inc. (Unknown); BJC HealthCare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202401096; 24FIM1268045 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Food Insecurity

STUDY DESIGN:
Intervention Model Description: 240 patients will be randomized to three arms: "usual care," NutriConnect Credit, and NutriConnect Delivery with equivalent monetary value to credit. The interventions will last 6 months.
Who Masked: Outcomes Assessor
Masking Description: Due to the open study design, the NutriConnect team will not be able to have either patient or research coordinator/Schnucks intervention delivers blinded on group assignment. However, the assignment will be hidden from research faculty, the study biostatistician, and study analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Control) (No Intervention): Patient is screened for food or financial insecurity, if positive, social worker will refer him/her to community service programs.
- NutriConnect Credit (Experimental): Patient is given $20 credit to their Schnucks (grocery) Reward account every other week for F&V shopping.
  Interventions: Other: Product prescription program- NutriConnect Credit
- NutriConnect Delivery (Experimental): Patient receives produce (F&V) box (with equivalent $20 value) delivered to home every other week.
  Interventions: Other: Product prescription program- NutriConnect Delivery

INTERVENTIONS:
Other: Product prescription program- NutriConnect Credit — Patient is given $20 credit to their Schnucks (grocery) Rewards account every other week for F&V shopping. The Rewards credit can be used either through the Schnucks App or in store.
  Arms: NutriConnect Credit
Other: Product prescription program- NutriConnect Delivery — Patient receives produce (F&V) box (equivalent $20 value) delivered to home every other week. The items in the box will be pre-selected by Schnucks and the NutriConnect dieticians.
  Arms: NutriConnect Delivery

SUMMARY:
The produce prescription program is one type of food is medicine (FIM) programs, where healthcare providers "prescribe" fruits and vegetables (F&V) to patients with low household incomes, experience food insecurity, and one or more diet-related diseases. NutriConnect seeks to compare the effectiveness of two produce prescription approaches on F&V intake and food security: credit to Rewards account (NutriConnect Credit) vs. produce box delivery (NutriConnect Delivery), while exploring implementation outcomes such as reach, sustainability, implementation, and cost.

DETAILED DESCRIPTION:
The Produce Prescription Program, as one type of Food is Medicine (FIM) initiatives, involves healthcare providers prescribing fruits and vegetables to patients often have low incomes, food insecurity, and diet-related illnesses. Previous systematic reviews have shown that these programs are associated with increased consumption of fruits and vegetables, improved diet quality, reduced food insecurity, and better management of diet-related diseases. However, the diversity in study designs, small sample sizes, and varied intervention intensities have limited the conclusive understanding of the full effects of these programs. Despite their potential benefits, critical gaps persist, notably in identifying the most effective strategies for socioeconomically disadvantaged patients. Additionally, challenges surrounding scalability, implementation, and sustainability hinder the widespread adoption of these programs.

To address these gaps, the NutriConnect team employs a Designing for Dissemination and Sustainability (D4DS) approach informed by the PRISM/RE-AIM framework. This involves early engagement of key partners crucial for scalability and sustainability. The study team initiated a collaborative consortium comprising Washington University in St. Louis, BJC Healthcare, and Schnucks (regional grocery chain). NutriConnect integrates multilevel, multicomponent intervention components, including in-hospital social needs screening, produce prescription, grocery rewards, and a health and wellness program, all aimed at promoting better nutrition and health in the community. NutriConnect seeks to compare the effectiveness of two produce prescription approaches on fruits and vegetables intake and food security: credit to Rewards account (NutriConnect Credit) vs. produce box delivery (NutriConnect Delivery), while exploring implementation outcomes, with the following aims.

Aim 1. Evaluate and compare the effectiveness of NutriConnect Credit with NutriConnect Delivery on changes in fruit and vegetable intake, food security, and self-reported health status.

Aim 2. Explore the scalability, sustainability, and determinants of the NutriConnect program guided by PRISM/RE-AIM, aiming to identify factors crucial for future scale-up.

Aim 3. Determine the implementation costs of NutriConnect using time-driven activity-based costing approach.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>= 18 years)
2. Received care at either medical floors or observation unit at the Bares Jewish Hospital (BJH), and discharged to home.
3. Being screened positive for food or financial insecurity.
4. Have elevated cardiovascular risk, i.e., self-reported diabetes, hypertension, hyperglycemia, or calculated BMI meeting obesity.

Exclusion Criteria:

1. Does not have competence to provide informed consent.
2. Is under suicide watch.
3. Is in police custody.
4. In hospice or palliative care.
5. Not have a stable home.
6. Is pregnant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
change in F&V intake | 6-month
  pre- and post-changes in F&V consumption (cups/day, continuous).

SECONDARY OUTCOMES:
Household food insecurity | 6-month
  pre- and post-changes in household food insecurity (binary). 6-item USDA Food Security Survey, minimum value = 0, maximum value = 6, lower the score means higher the food security

OTHER OUTCOMES:
Self-reported health status | 6-month
  pre- and post-changes in self-reported health status (5-point Likert scale, ordinal). 5-point Likert Scale: minimum value = 1, maximum value= 5, higher score means better outcome (or strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, MD, DrPH, MS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The data includes self-reported socio-demographic information, data on fruit and vegetable intake, food security status, and health status. Qualitative data includes implementation process, experiences and perspectives of both the intervention delivers and recipients, and other implementation-related factors and outcomes. The dataset includes de-identified quantitative data sets, transcriptions of qualitative interviews, codebooks for all qualitative and quantitative data, descriptive documentation of variables along with their relationships to outcomes, as well as the analytic plan and program.
  For the purposes of sharing and disseminating, all direct identifiers and any indirect identifiers that could be used in conjunction with other publicly available information to identify individuals will be removed from the study data. All transcriptions of focus group will also be void of any personal identifiers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available after 06/30/2025, and for 2 years.
Access Criteria: research protocol review and approval

REFERENCES:
- [Derived] Yoo SGK, Tabak RG, Mazzucca-Ragan S, Primo A, Bohannon D, Hashimoto D, Goss CW, Wu JH, Eromosele E, Hassanieh I, Hively A, Martinez A, Wang J, Huffman MD, Li J. NutriConnect: Enhancing health and food security through sustainable solutions and partnerships: Design and protocol of a pragmatic comparative effectiveness trial. Contemp Clin Trials. 2025 Nov;158:108083. doi: 10.1016/j.cct.2025.108083. Epub 2025 Sep 17. PMID 40972889